CLINICAL TRIAL: NCT06118151
Title: A Phase I, Parallel, Randomized, Active-controlled, Multi-center, Dose-escalation Study With Early Safety Data Reviews to Assess Safety and Immunogenicity of a Monovalent mRNA Vaccine Encoding Influenza Hemagglutinin in Adults 18 Years of Age and Older
Brief Title: Safety and Immunogenicity of a Monovalent mRNA Vaccine Encoding Influenza Hemagglutinin in Adult Participants 18 Years of Age and Older
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAV00018; U1111-1271-2001 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Influenza; Influenza Immunization
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Open label (Sponsor) Blinded (Sites, except for those preparing/administering study intervention)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- sentinel cohort 1 (Experimental): 20 Participants in each age group will receive either Influenza hemagglutinin mRNA vaccine candidate dose 1 or dose 2 and half number of the participants in each age group also receiving the RIV4 control
  Interventions: Biological: Influenza Hemagglutinin mRNA vaccine; Biological: Quadrivalent Recombinant Influenza Vaccine
- sentinel cohort 2 (Experimental): 20 Participants in each age group will receive either Influenza hemagglutinin mRNA vaccine candidate dose 3 or dose 4 and half number of the participants in each age group also receiving the RIV4 control
  Interventions: Biological: Influenza Hemagglutinin mRNA vaccine; Biological: Quadrivalent Recombinant Influenza Vaccine
- sentinel cohort 3 (Experimental): 10 Participants in each age group will receive Influenza hemagglutinin mRNA vaccine candidate dose 5 with half of the participants in each age group also receiving the RIV4 control
  Interventions: Biological: Influenza Hemagglutinin mRNA vaccine; Biological: Quadrivalent Recombinant Influenza Vaccine
- main cohort 1 (Experimental): 40 Participants in each age group will receive either Influenza hemagglutinin mRNA vaccine candidate dose 1 or dose 2 and half number of the participants in each age group also receiving the RIV4 control
  Interventions: Biological: Influenza Hemagglutinin mRNA vaccine; Biological: Quadrivalent Recombinant Influenza Vaccine
- main cohort 2 (Experimental): 40 Participants in each age group will receive either Influenza hemagglutinin mRNA vaccine candidate dose 3 or dose 4 and half number of the participants in each age group also receiving the RIV4 control
  Interventions: Biological: Influenza Hemagglutinin mRNA vaccine; Biological: Quadrivalent Recombinant Influenza Vaccine
- main cohort 3 (Experimental): 20 Participants in each age group will receive Influenza hemagglutinin mRNA vaccine candidate dose 5, and half number of the participants in each age group also receiving the RIV4 control
  Interventions: Biological: Influenza Hemagglutinin mRNA vaccine; Biological: Quadrivalent Recombinant Influenza Vaccine

INTERVENTIONS:
Biological: Influenza Hemagglutinin mRNA vaccine — Pharmaceutical form:Solution for injection-Route of administration:IM injection
Biological: Quadrivalent Recombinant Influenza Vaccine — Pharmaceutical form:Solution for injection-Route of administration:IM injection
  Other Names: RIV4; Flublok Quadrivalent®

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of a single intramuscular (IM) injection of different dose levels of messenger ribonucleic acid (mRNA) vaccine encoding influenza hemagglutinin compared to an active control quadrivalent recombinant influenza vaccine (RIV4) in adults 18 years of age and older. Study details include:

Study Duration: approximately 6 months Treatment Duration: 1 injection of mRNA vaccine encoding influenza hemagglutinin encoding influenza hemagglutinin or control.

Visit Frequency: Screening visit, Day 01, Day 02, Day 03, Day 09, Day 29, Day 91, Day 181

DETAILED DESCRIPTION:
Approximately 6 months

ELIGIBILITY:
Inclusion Criteria:

* Having given written informed consent prior to undertaking any study-related procedure. Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:
* Any subject who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Presence of any unsolicited systemic adverse events (AEs) reported in the 30 minutes after injection | Within 30 minutes after injection
  Number of participants with unsolicited systemic immediate adverse events (AEs)
Presence of solicited injection site reactions (ie, pre listed in the participant's diary card [DC] and in the electronic case report form [eCRF]) occurring up to 7 days after injection | Up to 7 days after injection
  Number of participants with solicited injection site reactions
Presence of solicited systemic reactions (ie, pre-listed in the participant's DC and in the eCRF) occurring up to 7 days after injection | Up to 7 days after injection
  Number of participants with solicited systemic reactions
Presence of unsolicited AEs reported up to 28 days after injection | Up to 28 days after injection
  Number of participants with unsolicited AEs
Presence of medically attended AEs (MAAEs) reported up to 28 days after injection | Up to 28 days after injection
  Number of participants with medically attended adverse events (MAAE)s
Presence of serious adverse events (SAEs) and adverse events of special interest (AESIs) throughout the study | From baseline up to 6 months
  Number of participants with serious adverse events (SAEs)
Presence of out-of-range biological test results (including shift from baseline values) up to 28 days after injection | Up to 28 days after injection
  Number of participants with out-of-range biological test results

SECONDARY OUTCOMES:
Hemagglutination inhibition (HAI) antibody (Ab) titers to homologous H3 strain at D29, D91, and D181 | At Day 29, Day 91, and Day 181
  Antibody titers are expressed as Geometric Mean Titers (GMTs)
Individual HAI Ab titer ratio D29/D01, D91/D01, D91/D29, D181/D01, and D181/D29 | From baseline up to 6 months
  Ratios of antibody titers measured by HAI in each group before and after vaccination
HAI Ab titer ≥ 40 [1/dil] at D29, D91, and D181 | At Day 29, Day 91 and Day 181
2-fold and 4-fold rise in HAI titers from D01 to D91 and D01 to D181 | From Day 01 through Day 91 and Day 01 through Day 181
Neutralizing Ab titers to homologous H3 strain at D29, D91, and D181 | At Day 29, Day 91, and Day 181
Individual neutralizing Ab titer ratio D29/D01, D91/D01, D91/D29, D181/D01, and D181/D29 | From baseline up to 6 months
2-fold and 4-fold rise in neutralizing titers from D01 to D91 and D01 to D181 | From Day 01 through Day 29 and Day 01 through Day 181
HAI Ab titers to selected heterologous H3 strains at D01, D29, D91, and D181 | At Day 01, Day 29, D91 and D181
Neutralizing Ab titers to selected heterologous H3 strains at D01, D29, D91, and D181 | At Day 01, Day 29, Day 91, and Day 181

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Peninsula Research Associates Site Number : 8400013, Rolling Hills Estates, California
  - Optimal Research Site Number : 8400026, San Diego, California
  - AMR Coral Gables/Miami, Formerly Clinical Research of South Florida, an AMR company (Clinic) Site Number : 8400004, Coral Gables, Florida
  - Research Centers of America Site Number : 8400003, Hollywood, Florida
  - Meridian Clinical Research, LLC Site Number : 8400016, Savannah, Georgia
  - AES Peoria Site Number : 8400017, Peoria, Illinois
  - AMR El Dorado Site Number : 8400009, El Dorado, Kansas
  - AMR - Newton Site Number : 8400005, Newton, Kansas
  - AMR Wichita West Site Number : 8400030, Wichita, Kansas
  - AMR Lexington Site Number : 8400014, Lexington, Kentucky
  - Benchmark Research Site Number : 8400010, Metairie, Louisiana
  - Quality Clinical Research Site Number : 8400018, Omaha, Nebraska
  - Velocity Clinical Research, Omaha Site Number : 8400007, Omaha, Nebraska
  - Velocity Clinical Research Vestal Site Number : 8400033, Vestal, New York
  - Coastal Carolina Research Center - N Charleston Site Number : 8400008, North Charleston, South Carolina
  - AMR Knoxville Site Number : 8400027, Knoxville, Tennessee
  - Elligo Health Research, Inc. Site Number : 8400035, Austin, Texas
  - Benchmark Research - Austin Site Number : 8400006, Austin, Texas
  - AES Austin Site Number : 8400021, Austin, Texas
  - Clinical Trials of Texas, Inc. Site Number : 8400012, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org